CLINICAL TRIAL: NCT05234892
Title: ALTo endogrAft Italian Registry
Acronym: ALTAIR
Status: Recruiting | Type: Observational
Sponsor: Gianmarco de Donato (Other)
Collaborators: University of Roma La Sapienza (Other); University of Siena (Other)
Responsible Party: Sponsor-Investigator, Gianmarco de Donato, Associate Professor, Azienda Ospedaliera Universitaria Senese
Organization: Azienda Ospedaliera Universitaria Senese (Other)
Other Study IDs: ALTAIR001
Record Dates: First submitted 2022-01-28; First posted 2022-02-10 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm; AAA; Endovascular Aneurysm Repair; EVAR; Endograft
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- EVAR group: All consecutive eligible patients submitted to EVAR by Alto Endovascular AAA implantation will be included in analysis. Patients will be submitted to EVAR procedures on the basis of their own preferences, anatomical features, and operators experience.
  Interventions: Device: ALTO endograft implantation

INTERVENTIONS:
Device: ALTO endograft implantation — Implantantion of aorto-bisiliac ALTO endograft to exclude Abdominal Aortic Aneurysms

SUMMARY:
The aim of present study is to evaluate intraoperative, peri-operative, and post-operative results in patients treated by the ALTO stent graft (Endologix Inc. Irvine, Calif) for elective Abdominal Aortic Aneurysm repair in a multicentric consecutive experience.

DETAILED DESCRIPTION:
Thirty years ago, Juan Parodi developed the first prototype of endograft for Endovascular Aneurysm Repair, a handmade device made of a tube-shaped aorto-aortic graft sutured at each end to a balloon-expandable stent based on the design of radiologist Julio Palmaz. This device was implanted in a human body for the first time on September 7, 1990, in Buenos Aires, Argentina. By 1994, the first commercially available devices had been launched onto the market. Stent-graft material and design changed in various ways to improve conformability, reduce fracture, and minimize device migration rates. Over the years Endovascular Aneurysm Repair has become an effective treatment of AAA in challenging anatomy as hostile neck and small access. These performances have been achieved thanks to continuous technological development to overcome the previous limitation in Endovascular Aneurysm Repair applicability. Since 2010, the Ovation Abdominal Stent Graft System (Endologix Inc. Irvine, Calif) has offered a new concept of sealing, achieved by a network of O-rings filled with a polymer that can treat a great variety of difficult anatomies through a low-profile platform. In the latest version of the stent-graft, called Ovation Alto, the conformable O-rings with CustomSealTM polymer have been repositioned near the top of the endograft, providing a seal just below the renal arteries. Very few papers were published highlighting the early and late outcomes of this new device. In this perspective, this study is intended to be the first multicenter prospective registry regarding the implantation of Alto stent graft.

ELIGIBILITY:
Inclusion Criteria:

* Elective AAA patients that should be treated by standard EVAR, according to Endologix Alto endograft device's Instructions For Use;
* Patient is willing to comply with specified follow-up evaluations at the specified times for the duration of the study;
* Patient is >18 years old;
* Patient, or their legal representative, understands the nature of the procedure and provides written informed consent, prior to enrollment in the study.

Exclusion Criteria:

* EVAR performed in Urgent/Emergent setting;
* Patients treated outside Endologix Alto endograft device's Instructions For Use;
* Patients refusing treatment;
* Patients for whom antiplatelet therapy, anticoagulants or antihypertensive drug are contraindicated;
* Patients with a history of prior life-threatening contrast medium reaction;
* Life expectancy of less than follow-up period.

AAA: abdominal aortic aneurysm; EVAR: abdominal endovascular aneurysm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive eligible patients submitted to EVAR by Alto Endovascular AAA implantation will be included in analysis. Patients will be submitted to EVAR procedures on the basis of their own preferences, anatomical features, and operators experience.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical success | 90 days
  correct graft deployment without any unintentional occlusion of the aortic visceral branches and/or both hypogastric arteries, with aneurysm exclusion confirmed by the intraoperative angiography, without signs of type I/III endoleak a conversion to open surgery.
Technical success | 1 year
  correct graft deployment without any unintentional occlusion of the aortic visceral branches and/or both hypogastric arteries, with aneurysm exclusion confirmed by the intraoperative angiography, without signs of type I/III endoleak a conversion to open surgery.
Technical success | 5 years
  correct graft deployment without any unintentional occlusion of the aortic visceral branches and/or both hypogastric arteries, with aneurysm exclusion confirmed by the intraoperative angiography, without signs of type I/III endoleak a conversion to open surgery.
Clinical success | 90 days
  Successful deployment of the endovascular device at the intended location without death as a result of aneurysm-related treatment, type I or III endoleak, or graft infection or thrombosis, aneurysm expansion (>5 mm), aneurysm rupture, or conversion to open repair. Moreover, the presence of graft dilatation of 20% or more by diameter, graft migration, or a failure of device integrity.
Clinical success | 1 year
  Successful deployment of the endovascular device at the intended location without death as a result of aneurysm-related treatment, type I or III endoleak, or graft infection or thrombosis, aneurysm expansion (>5 mm), aneurysm rupture, or conversion to open repair. Moreover, the presence of graft dilatation of 20% or more by diameter, graft migration, or a failure of device integrity.
Clinical success | 5 years
  Successful deployment of the endovascular device at the intended location without death as a result of aneurysm-related treatment, type I or III endoleak, or graft infection or thrombosis, aneurysm expansion (>5 mm), aneurysm rupture, or conversion to open repair. Moreover, the presence of graft dilatation of 20% or more by diameter, graft migration, or a failure of device integrity.

SECONDARY OUTCOMES:
Operative time | Immediately after the procedure
  Duration of procedure
Radiation exposure | Immediately after the procedure
  Radiation exposure during endovascular procedure
Contrast medium usage | Immediately after the procedure
  Amount of contrast medium usage during procedure
Abdominal Aortic Aneurysm Shrinkage | 1 year
  AAA diameter reduction after EVAR
Abdominal Aortic Aneurysm Shrinkage | 5 year
  AAA diameter reduction after EVAR

CONTACTS AND LOCATIONS:
Overall Officials: Gianmarco de Donato, MD, PhD, Principal Investigator — University of Siena; Maurizio Taurino, MD, PhD, Principal Investigator — University La Sapienza of Rome; Francesco Talarico, MD, PhD, Principal Investigator — Ospedale Civico di Palermo
Locations (2):
- Italy (2):
  - University La Sapienza of Rome, Rome
  - University of Siena, Siena

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Donato G, Pasqui E, Panzano C, Brancaccio B, Grottola G, Galzerano G, Benevento D, Palasciano G. The Polymer-Based Technology in the Endovascular Treatment of Abdominal Aortic Aneurysms. Polymers (Basel). 2021 Apr 7;13(8):1196. doi: 10.3390/polym13081196. PMID 33917214
- [Result] de Donato G, Setacci F, Sirignano P, Galzerano G, Borrelli MP, di Marzo L, Setacci C. Ultra-low profile Ovation device: is it the definitive solution for EVAR? J Cardiovasc Surg (Torino). 2014 Feb;55(1):33-40. PMID 24356044
- [Result] de Donato G, Pasqui E, Panzano C, Galzerano G, Cappelli A, Palasciano G. Early Experience with the New Ovation Alto Stent Graft in Endovascular Abdominal Aortic Aneurysm Repair. EJVES Vasc Forum. 2021 Nov 27;54:7-12. doi: 10.1016/j.ejvsvf.2021.11.003. eCollection 2022. PMID 34950916
- [Result] Sirignano P, Mansour W, Capoccia L, Cuozzo S, Camparini S, de Donato G, Mangialardi N, Ronchey S, Talarico F, Setacci C, Speziale F; Collaborators. Endovascular aortic repair in patients with challenging anatomies: the EXTREME study. EuroIntervention. 2021 Apr 2;16(18):e1544-e1550. doi: 10.4244/EIJ-D-19-00547. PMID 31793884
- [Result] Holden A, Lyden S. Initial experience with polymer endovascular aneurysm repair using the Alto stent graft. J Vasc Surg Cases Innov Tech. 2020 Feb 1;6(1):6-11. doi: 10.1016/j.jvscit.2019.04.007. eCollection 2020 Mar. PMID 32025596
- [Result] Barleben A, Mathlouthi A, Mehta M, Nolte T, Valdes F, Malas MB; Ovation trial investigators. Long-term outcomes of the Ovation Stent Graft System investigational device exemption trial for endovascular abdominal aortic aneurysm repair. J Vasc Surg. 2020 Nov;72(5):1667-1673.e1. doi: 10.1016/j.jvs.2020.01.066. Epub 2020 Apr 2. PMID 32249041
- [Result] de Donato G, Pasqui E, Mele M, Panzano C, Giannace G, Setacci F, Benevento D, Setacci C, Palasciano G. The use of a low-profile stent graft with a polymer ring sealing technology combined with bare renal stent (vent technique) in patients with juxtarenal aneurysm not eligible for open surgery and fenestrated endograft. J Vasc Surg. 2020 Jun;71(6):1843-1850. doi: 10.1016/j.jvs.2019.06.220. Epub 2019 Oct 31. PMID 31676183
- [Derived] de Donato G, Pasqui E, Sirignano P, Talarico F, Palasciano G, Taurino M; ALTAIR collaborators. Endovascular Abdominal Aortic Aneurysm Repair With Ovation Alto Stent Graft: Protocol for the ALTAIR (ALTo endogrAft Italian Registry) Study. JMIR Res Protoc. 2022 Jul 11;11(7):e36995. doi: 10.2196/36995. PMID 35816378